# Taking a Look at Patient Experiences In Rectal Cancer Clinical Trials

This is an informed consent form for rectal cancer patients joining <a href="Power Clinical Trial's">Power Clinical Trial's</a> observational medical trial.

Date: June 8, 2023

#### Introduction

Rectal cancer, also known as colorectal cancer, is a type of cancer that develops in the cells of the rectum, which is the final portion of the large intestine. The large intestine, or colon, connects the small intestine to the anus. Rectal cancer typically begins as small growths called polyps on the inner lining of the rectum. Over time, some of these polyps can become cancerous and develop into tumors.

Observational trials help identify risk factors associated with rectal cancer development, such as age, family history, lifestyle choices, and other environmental factors. By studying a large population over an extended period, researchers can analyze data to determine which factors increase the likelihood of developing rectal cancer.

We are studying why some people with rectal cancer may not want to join or finish other studies that test new treatments. We want you to be part of our study, where we will look at your medical records and ask you some questions. We want to know what makes you decide to join or not join other studies that test new treatments. We promise to keep your information private and use it only for this study.

This study is not about testing any new treatments but only about learning from you. Being in this study does not mean you will get any different treatment than what your doctor gives you. This paper will tell you everything you need to know about the survey, how to join it, and who will work with you.

# Identifying Challenges and Solutions to Improve Participation and Completion

The primary objective of this research study is to explore the barriers encountered by specific demographic groups of rectal cancer patients during their engagement in clinical trials, which historically lack diverse representation. We aim to collect comprehensive information from participants and identify common factors that impede their enrollment or successful completion of these trials.

By carefully analyzing data from various demographic perspectives, this study aims to uncover patterns that impact the experiences of future rectal cancer patients. Your active involvement in this crucial research is of utmost importance, as it can offer unique insights to enhance the participation and completion rates of rectal cancer patients in clinical trials.

#### What You Should Be Aware Of

Participation in this study is optional, and you can withdraw at any point without facing any consequences. It is important to emphasize that your decision to participate or decline will not affect how it treats you.

In medical research investigations, it is standard procedure to ensure voluntary participation. Additionally, this research is purely observational, which means that if you are already receiving treatment, your diagnosis, medication, and care will continue as usual. The study team prohibits interfering with your medical care or monitoring how it treats you.

Enrolling in an interventional clinical trial is imperative to participate in this research study on rectal cancer. It should emphasize that joining this observational clinical study will not interfere with your ongoing treatment plan for rectal cancer, even if you are already involved in a separate clinical trial.

If you have any inquiries regarding your participation or involvement, feel free to ask in the interventional clinical trial; seeking guidance from your healthcare team is strongly recommended. They can provide detailed information and address any concerns you may have. It is crucial to fully comprehend the disparities between interventional clinical trials and their implications.

#### Active Participation And Subsequent Phone Follow-up Conversations

Your full participation in this observational clinical study entails completing biweekly surveys within a 30-minute timeframe. Dedicated quarterly follow-up conversations are scheduled for your engagement in the interventional clinical trial. To actively participate in both research components, following the study's guidelines is of utmost importance by promptly organizing and attending these calls.

#### Precautionary Measures in the Research Investigation

When considering this observational clinical trial, it is imperative to highlight its associated risks. Since the study solely relies on observational methods, no changes will establish care regimens, unequivocally eliminating potential adverse effects on participants.

Furthermore, to ensure the utmost confidentiality, we have implemented robust encryption mechanisms and stringent password protection measures to strengthen the security of all electronic data. These rigorous safeguards effectively mitigate the risk of unauthorized access or breaches during customary video conferences and online reporting, thereby enhancing the overall framework for data protection.

## **Potential Advantages**

Careful assessment is essential for this rectal cancer clinical trial, as it holds considerable potential benefits. The trial's findings will provide invaluable insights into the factors that influence the enrollment and retention rates of a heterogeneous group of patients with rectal cancer in clinical studies.

This knowledge will serve as a vital foundation for improving subsequent clinical trials that aim to include individuals with rectal cancer. By actively participating in this study, you can make a substantial and meaningful contribution to advancing our understanding of the factors that may impact the involvement of diverse patient populations in rectal cancer trials.

#### This Study Versus Other Rectal Cancer Clinical Trials

Unlike numerous other investigations on rectal cancer, this study adopts a unique observational approach. In this study, participants are not obliged to adhere to any predetermined treatment plan.

Although the research team may not possess all knowledge about rectal cancer studies, resources are available to support you. ClinicalTrials.gov presents a comprehensive inventory of <u>rectal cancer studies</u>, and Power's reference page compiles the latest information on ongoing <u>rectal cancer clinical trials</u> actively seeking volunteers.

#### Exploring Inclusivity in Clinical Trials: Suggested Resources

Despite the limited examination of diverse populations' presence in clinical trials, several studies present valuable perspectives. Below, we present a compilation of suggested readings that are both captivating and informative:

Mak, Winnie WS, Rita W. Law, Jennifer Alvidrez, and Eliseo J. Pérez-Stable. "Gender and ethnic diversity in NIMH-funded clinical trials: Review of a decade of published research." Administration and Policy in Mental Health and Mental Health Services Research 34 (2007): 497-503.

<u>Varma, Tanvee, Camara P. Jones, Carol Oladele, and Jennifer Miller. "Diversity in clinical research: public health and social justice imperatives." *Journal of Medical Ethics* 49, no. 3 (2023): 200-203.</u>

These readings provide valuable insights into involving diverse populations in clinical trials and understanding the importance of inclusivity in research.

## **Protecting Your Privacy Effectively**

We take your privacy seriously in this clinical study and have implemented strict measures to protect it. Your records have assigned a unique code or number for complete anonymity throughout the study. All identifying materials are securely stored under the close supervision of the researcher in a locked file cabinet. We highly value your privacy and attempt not to disclose personal information without your explicit consent, except when required by law.

Verification Of Voluntary Involvement And Consent.

By affixing my signature below, I confirm that I have received comprehensive details regarding the nature and objectives of this study. My involvement in this study is entirely voluntary, and I retain the freedom to withdraw my participation at any time without encountering any adverse repercussions.

I understand that the decision to withdraw will not impact my present or future medical care. Furthermore, I request a copy of this consent form for my records.

| Printed Name of Participant |
|-----------------------------|
| Signature |
| <br>Date |

Verification of Participant's Understanding

As the clinical trial personnel responsible for discussing the consent form with the participant, I am delighted to confirm that the participant has exhibited an understanding of the risks, benefits, and procedures associated with this clinical research.

Through transparent and informative discussions, all questions and uncertainties have been thoroughly addressed, ensuring that the participant has a clear comprehension of the implications and protocols of the study.

| Printed Name of Person Getting Consent |
|----------------------------------------|
| Signature of Person Getting Consent |
| <br>Date |